CLINICAL TRIAL: NCT04738903
Title: Q Value Customized Versus Wavefront Optimized Ablation in Femtosecond Laser-Assisted LASIK for Myopia and Myopic Astigmatism. A Contralateral Comparative Study
Brief Title: Q Value Customized Versus Wavefront Optimized Ablation in Femtosecond Laser-Assisted LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Principal Investigator, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CQLASIK
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Patients With Myopic Spherical Equivalent up to -12 Diopters
Keywords: Femtosecond LASIK; Q value; Wave-front Optimized (WFO)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom Q treatment group (Active Comparator): For every patient, the eye with the greater myopic spherical equivalent (SE) will be assigned for the Custom-Q treatment group.
  Interventions: Procedure: Femtosecond laser assisted LASIK eye surgery
- Wave-front optimized (WFO) group (Active Comparator): For every patient, the other eye with the lesser myopic SE will be assigned for the WFO treatment group
  Interventions: Procedure: Femtosecond laser assisted LASIK eye surgery

INTERVENTIONS:
Procedure: Femtosecond laser assisted LASIK eye surgery — FS-LASIK eye surgery includes corneal flap creation with femtosecond laser using the Femtosecond laser WaveLight FS200 followed by excimer laser vision correction of the patient's refractive error using excimer laser WaveLight EX500.

SUMMARY:
Corneal asphericity is expressed numerically as the "Q-value". A minus value means that corneal curvature flattens towards the periphery and the cornea is prolate in shape, but when the curvature steepens towards the periphery, the cornea is oblate in shape and has a positive Q-value.

The current study evaluates the effect of LASIK eye surgery on corneal asphericity by comparing 2 software treatment platforms; the Q value customized ablation versus the conventional Wave-front optimized ablation in a fellow eye study pattern.

DETAILED DESCRIPTION:
The standard excimer laser correction of myopia is associated with decreased visual quality in the form of a decrease in contrast sensitivity and night vision. This degradation of the visual quality is attributed to changes in the corneal asphericity that increase the high order aberrations (HOAs), such as spherical aberrations because it leads to shifting of the corneal asphericity towards the oblate shape.

The wavefront-optimized (WFO) profile avoids the creation of new HOAs, but it is not able to treat those which are already present pre-operatively.

The Q-adjusted treatments correct the sphero-cylindrical refractive errors and try to maintain the corneal asphericity at the same time, but like the WFO ablation profiles, it is limited to correcting the spherical aberrations and not the non-rotational symmetric HOAs.

Some studies compared Lasers of two different platforms on contralateral eyes of the same patient in order to minimize inter-patient differences such as corneal wound healing and corneal biomechanics. By exclusion of these inter-patient differences, a more accurate judgment on the outcomes can be achieved.

ELIGIBILITY:
Inclusion Criteria: Candidates for Laser vision correction (LVC) with

1. Myopic Spherical Equivalent up to -12 diopters.
2. Myopic astigmatism up to -6 diopters.
3. Corneal thinnest location ≥ 500 um 4- Residual stromal bed ≥ 300 um.

Exclusion Criteria:

1. Patients not candidates for LVC.
2. Hyperopic patients or mixed astigmatism.
3. Systemic disease that contraindicates LVC.
4. Intra- or post-operative complications. 5- Previous corneal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Q value | 6 months
  Pentacam evaluation of post-LASIK Q value

SECONDARY OUTCOMES:
Postoperative corneal thickness at the pupillary center | 6 months
  Pentacam evaluation of post-LASIK pachymetry at the pupil center

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdel-Radi, MD, Principal Investigator — Assiut University
Locations (1):
- TIBA eye center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piao J, Li YJ, Whang WJ, Choi M, Kang MJ, Lee JH, Yoon G, Joo CK. Comparative evaluation of visual outcomes and corneal asphericity after laser-assisted in situ keratomileusis with the six-dimension Amaris excimer laser system. PLoS One. 2017 Feb 10;12(2):e0171851. doi: 10.1371/journal.pone.0171851. eCollection 2017. PMID 28187180
- [Derived] Mostafa MM, Abdelmotaal H, Abdelazeem K, Goda I, Abdel-Radi M. Q-value customized versus wavefront-optimized ablation in femtosecond laser-assisted LASIK for myopia and myopic astigmatism: a prospective contralateral comparative study. Eye Vis (Lond). 2022 Nov 2;9(1):43. doi: 10.1186/s40662-022-00312-3. PMID 36320050